CLINICAL TRIAL: NCT01728441
Title: REAL PTX - Randomized Evaluation of the Zilver PTX Stent vs. Paclitaxel-Eluting Balloons for Treatment of Symptomatic Peripheral Artery Disease of the Femoropopliteal Artery
Brief Title: Evaluation of Paclitaxel Eluting Stent vs Paclitaxel Eluting Balloon Treating Peripheral Artery Disease of the Femoral Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Provascular GmbH (Other)
Collaborators: William Cook Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prov 01-2012; U1111-1136-8610 (Other: WHO)
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Peripheral Artery Disease
Keywords: PAD; stenting; angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel Eluting Stent (Experimental): Patients randomized to treatment with paclitaxel eluting stent will receive the Zilver® PTX® stent.Primary stenting should be performed covering the full lesion. Post-dilatation is at the investigator's discretion.
  Interventions: Device: Paclitaxel Eluting Stent
- Paclitaxel Eluting Balloon (Active Comparator): For patients randomized to treatment with drug eluting balloon (DEB), angioplasty (ballooning) should be performed covering the full lesion.
  Interventions: Device: Paclitaxel Eluting Balloon

INTERVENTIONS:
Device: Paclitaxel Eluting Stent
  Other Names: Zilver PTX stent
  Arms: Paclitaxel Eluting Stent
Device: Paclitaxel Eluting Balloon
  Arms: Paclitaxel Eluting Balloon

SUMMARY:
Objective of the REAL PTX trial is to compare paclitaxel-eluting stents to paclitaxel-eluting balloons for treating symptomatic peripheral artery disease of the femoropopliteal artery.

DETAILED DESCRIPTION:
The REAL PTX trial has been designed as prospective, randomized, multi-center, post-market study investigating the effect of the paclitaxel-eluting stent Zilver® PTX® (DES)in comparison to the use of a paclitaxel eluting balloon (DEB)in treating symptomatic peripheral artery disease of the femoropopliteal artery.

Up to 150 patients will be enrolled in Germany and Belgium. Enrollment is expected to be completed within approximately six months of initiating the study.

One group (DES or DEB) will be considered to yield significantly better results of the primary patency rate than the other group at 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥ 18
* Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form.
* Subject understands the duration of the study, agrees to attend follow-up visits, and agrees to complete the required testing.
* Rutherford category 2-5.
* Subject has a de novo or restenotic lesion with ≥ 70% stenosis documented angiographically and no prior stent in the target lesion.
* Target lesion is at least 1cm below the origin of the profunda femoris and does not exceed the medial femoral epicondyle.
* A single target lesion (stenotic areas separated by more than 3 cm with ≤ 30% stenosis might, at the decision of the investigator, be considered as 2 lesions).
* Reference vessel diameter (RVD) ≥ 4 mm and ≤ 6.5 mm by visual assessment.
* Patency of at least one (1) infrapopliteal artery to the ankle (< 50% diameter stenosis) in continuity with the native femoropopliteal artery.
* A guidewire has successfully traversed the target treatment segment.

Exclusion Criteria:

Clinical exclusion criteria

* Inability to obtain informed consent.
* Life expectancy < 12 months.
* Pregnancy, suspected pregnancy, or breastfeeding during study period (patients of childbearing potential must have negative serum pregnancy test 7 days prior to treatment).
* Presence of one or more of the following co-morbid factors: hemodialysis dependence, renal insufficiency with a serum creatinine ≥ 2.5 mg/dl, cerebrovascular accident (CVA) within 1 month of procedure or any CVA resulting in unresolved walking impairment, and/or myocardial infarction (MI) within 1 month of procedure.
* Any evidence of hemodynamic instability prior to procedure/randomization.
* Coagulopathy or clotting disorders.
* Present or suspected systemic infection or osteomyelitis affecting target limb.
* Contraindication to contrast media or any study-required medication (antiplatelets, anticoagulants, thrombolytics, etc).
* Hypersensitivity to nitinol and/or paclitaxel.
* Enrollment into another study.
* Intervention of the target lesion less than 90 days prior of the study procedure.

Anatomic Exclusion Criteria:

* Untreated external iliac artery inflow lesion (study allows for successful treatment prior to study treatment procedures).
* Total occlusion uncrossable by a conventional guidewire.
* Acute occlusive intraluminal thrombosis of the proposed lesion site.
* Evidence of an aneurysm at the target lesion site.
* Perforation in the target vessel as evidenced by the extravasation of contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity Ratio (PSVR) | 12 months
  The primary outcome will be the one-year primary patency rate (Kaplan-Meier estimate at 12 months).Primary patency is defined as absence of clinically-driven target lesion revascularization (TLR) or binary restenosis. Binary restenosis is defined as a peak systolic velocity ratio (PSVR) > 2.4 as evaluated by duplex ultrasound core laboratory analysis.
target lesion revascularization (TLR) | 12 months
  The primary outcome will be the one-year primary patency rate (Kaplan-Meier estimate at 12 months).Primary patency is defined as absence of clinically-driven target lesion revascularization (TLR) or binary restenosis. Binary restenosis is defined as a peak systolic velocity ratio (PSVR) > 2.4 as evaluated by duplex ultrasound core laboratory analysis.

SECONDARY OUTCOMES:
Major Adverse Events (MAEs) | 6, 12 and 24 months
  MAE is defined as:
  * Death within 30 days of the index procedure or within 30 days of a target lesion revascularization (TLR)
  * Clinically-driven TLR, or
  * Major target limb amputation.
All cause death | 6, 12 and 24 months
Target vessel revascularization (TVR) | 6, 12 and 24 months
Clinically-driven target lesion revascularization (TLR) | 6, 12 and 24 months
  Clinically-driven TLR is defined as a reintervention performed for ≥ 50% diameter stenosis (confirmed by angiography) within ± 5 mm proximal and/or distal to the target lesion after documentation of recurrent clinical symptoms of peripheral artery disease (PAD) following the initial procedure.
Major target limb amputation within 6, 12 and 24 months. Major target limb Major target limb amputation | 6, 12 and 24 months
  Major target limb amputation is defined as amputation of the target leg other than amputation of the toe(s).
Sustained clinical improvement | 6, 12 and 24 months
  Sustained clinical improvement is defined as an improvement in the Rutherford category of one class compared to baseline in surviving patients who are free from major target limb amputation and free from target lesion revascularization (TLR).
Binary restenosis | 6, 12 and 24 months
  Binary restenosis (Peak Systolic Velocity Ratio (PSVR) >2.4)of the target lesion at 6, 12 and 24 months or at the time of reintervention prior to any pre-specified time point.
Walking capacity | 6, 12 and 24 months
  Walking capacity assessment by walking impairment questionnaire (WIQ) at 6, 12 and 24 months or at the time of reintervention prior to any pre-specified time point.
Procedural success | 6, 12 and 24 months
  Procedural success is defined as obtainment of < 30% residual stenosis on angiography by visual estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Park Hospital Leipzig
Locations (5):
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius Department of Vascular Surgery, Dendermonde
- Germany (3):
  - Universitäts Herzzentrum Freiburg Bad Krozingen Abteilung Angiologie, Bad Krozingen
  - Angiologikum Hamburg Centre for Interventional Vascular Medicine, Hamburg
  - Park-Krankenhaus Leipzig, Leipzig

REFERENCES:
- [Derived] Bausback Y, Wittig T, Schmidt A, Zeller T, Bosiers M, Peeters P, Brucks S, Lottes AE, Scheinert D, Steiner S. Drug-Eluting Stent Versus Drug-Coated Balloon Revascularization in Patients With Femoropopliteal Arterial Disease. J Am Coll Cardiol. 2019 Feb 19;73(6):667-679. doi: 10.1016/j.jacc.2018.11.039. PMID 30765033